CLINICAL TRIAL: NCT02536716
Title: The Effect of Platform-Matching Versus Platform-Switching Using Standard Internal Versus Tapered Internal Plus Dental Implants on Peri-implant Hard and Soft Tissue Healing
Brief Title: The Effect of Platform-Matching Versus Platform-Switching Dental Implants on Peri-implant Hard and Soft Tissue Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Graduate Periodontics Program Director, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.0448
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Missing Tooth
Keywords: Dental Implant
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platform-matched dental implant (Active Comparator): Platform-matched dental implant placement to measure marginal bone loss, gingival margin position, and papilla fill.
  Interventions: Procedure: Platform-matched dental implant
- Platform-switched dental implant (Experimental): Platform-switched dental implant placement to measure marginal bone loss, gingival margin position, and papilla fill.
  Interventions: Procedure: Platform-switched dental implant

INTERVENTIONS:
Procedure: Platform-matched dental implant — A platform-matched dental implant will be placed surgically, restored with a crown and evaluated for up to 12 months.
  Arms: Platform-matched dental implant
Procedure: Platform-switched dental implant — A platform-switched dental implant will be placed surgically, restored with a crown and evaluated for up to 12 months.
  Arms: Platform-switched dental implant

SUMMARY:
To compare platform-switched implants to platform-matched implants for replacement of a single missing tooth and their effect on: 1) Interproximal alveolar crest level in relation to implant platform. 2) Buccal implant recession. 3) Presence or absence of black triangle apical to the contact point. 4) Implant Success. 5) Adequate buccal tissue thickness.

DETAILED DESCRIPTION:
Thirty patients will have a dental implant placed. Fifteen patients will be randomly selected by a coin toss to receive a platform-switched implant while the other fifteen will receive platform-matched implant. Each patient will receive a diagnostic work-up including standardized radiographs (periapicals), study casts, clinical photographs, and a clinical examination of teeth adjacent to the edentulous sites. Pre-surgical preparation will include detailed oral hygiene instructions. Baseline data will be collected at initial exam, and at 2, 4, 6, and 12 months. Parameters measured will include: plaque index, gingival index, probing depth, keratinized tissue, bleeding on probing, and digital radiographic examination. Pre-surgical measurements will include: cemento-enamel junction to osseous crest on adjacent teeth by direct measurement at surgery, and by radiograph at baseline, 2, 4, 6, and 12 months, periodontal form, periodontal biotype, tooth shape, and papilla harmony. Patients will be randomly selected for treatment group assignment using a coin toss before surgery by the mentor. One investigator who is unaware of group assignment will perform all baseline examinations and all follow-up examinations. Means and standard deviations will be calculated for all parameters. A paired t-test will be used to evaluate the statistical significance of the differences between initial and final data. An unpaired t-test will be used to evaluate statistical differences between the test and control groups. A sample size of 15 gives 80% statistical power to detect a difference of 0.5 mm of implant bone loss between groups. All surgical procedures will be completed by one operator under the direction of one mentor. Pre-surgical measurements will be taken first. Local anesthesia will be administered. The surgical procedure will consist of the reflection of full thickness flaps to expose the alveolar crest. The implant platform will be placed 3 to 4 mm apical to the mid-facial gingival margin using dental implant osteotomy drills for preparation of the site. The surgical procedures will be documented with clinical photographs. Sutures will be used to close the flap and bury the implant under the tissue. Records will be kept of healing periodically for the first 8 weeks, then at 4, 6 and 12 months. The test group will use a BioHorizons Tapered Internal Plus "platform-switched" implant. The control group will be BioHorizons standard Internal "platform-matched" implant. All patients will be seen at 1-2, 4, 6 and 8 weeks to monitor healing. At week 8 the implant will be uncovered surgically and provisionalized, and at the 4 month visit the final crown will be placed. Subsequent examinations will take place at 6 and 12 months. Post-surgically, patients will take an antibiotic (doxycycline hyclate 100 mg once a day for two weeks), an analgesic (Vicodin ES every 4-6 hours as needed for pain), and an anti-inflammatory agent (Naproxen 375mg every 12 hours for one week). At post-operative visits plaque removal, and oral hygiene instruction, as needed, will be performed along with clinical photographs and standardized radiographs as scheduled. The results of this study will allow comparison of peri-implant soft and hard tissue healing following placement of a BioHorizons "platform-switched" Tapered Internal Plus implant versus a standard Internal "platform-matched" implant in terms of the effect on marginal bone loss, buccal recession, and papilla fill.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have one edentulous site bordered by 2 teeth.
* 2. Healthy persons at least 18 years old.
* 3. Understands and has signed the informed consent.

Exclusion Criteria:

* 1. Patients with uncontrolled diabetes, immune disease, or systemic disease that significantly affects the periodontium.
* 2. Previous head and neck radiation.
* 3. Patients who have been on IV bisphosphonates or oral bisphosphonates for > 3 years.
* 4. Smokers.
* 5. Patients who need prophylactic antibiotics prior to dental procedures.
* 6. Patients with allergy to any medication or material used in the study.
* 7. Chemotherapy in the previous 12 months.
* 8. Severe psychological problems.
* 9. Patients unable to sign the informed consent.
* 10. Pregnant patients.
* 11. History of allergy to common dentifrice ingredients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Marginal alveolar bone loss | 12-months post dental implant placement
  Bone loss will be measured radiographically using a stent

SECONDARY OUTCOMES:
Buccal implant recession | 12-months post dental implant placement
  Buccal implant recession will be measured using a North Carolina probe using the adjacent teeth and incisal edge of the crown
Papilla fill | 12-months post dental implant placement
  Presence or absence of black triangle apical to the contact point
Buccal soft tissue thickness around implant | 12-months post dental implant placement
  Thickness will be measured with an endodontic file using a rubber stopper (objective measure of tissue thickness by penetrating tissue and measuring the thickness in mm).

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States